CLINICAL TRIAL: NCT01504009
Title: Investigating the Effect of Muscle Training in Patients With Amyotrophic Lateral Sclerosis and Looking Into the Mechanisms Behind Development of Muscle Atrophy
Brief Title: Muscle Training of Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALS-project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Line Jensen, PhD-student, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALS-2011.05
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Nervous System Disease; Neurodegenerative Disease; Motor Neuron Disease; ALS; Muscle training; Muscle atrophy
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Nervous System Diseases; Neurodegenerative Diseases; Motor Neuron Disease; Muscular Atrophy | interventions — Resistance Training; Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Muscle strength (Experimental)
  Interventions: Other: Muscle training

INTERVENTIONS:
Other: Muscle training — 12 weeks of strength training 2-3 times/week
  Other Names: Strength training; Rehabilitation

SUMMARY:
Patients with neuropathic diseases are experiencing increasing muscle weakness, loss of muscle strength and functional abilities during their illness. In healthy people, regular exercise is the best way to maintain or improve muscle strength, endurance and general health status and thereby maintain functioning abilities. Previously, patients with neuromuscular diseases were advised to avoid any kind of physical exercise. However, lately a number of studies have evaluated the effect of training in patients with neuromuscular diseases, and positive effects on the functional abilities have been found. Based on these findings we want to investigate the mechanisms leading to development of muscle atrophy and loss of functional abilities, and to explore the opportunities of reducing muscle wasting and thereby improve the course of the disease development through strength training.

The main objective is to investigate the effects of strength training on slowing disease progression and reduce the decline in muscle strength and function in patients with amyotrophic lateral sclerosis (ALS). In addition, the aim is to carry out detailed studies of biological processes in muscle tissue in order to unveil mechanisms leading to muscle atrophy, and to examine effects of a strength training program. The goal is to be able to incorporate strength training in the treatment program of these patients in order to maintain muscle strength and function in the individual for as long as possible.

Minimum 10 patients with the disease are included in the study. Through a 12 week period the patients will participate in strength training 2-3 times per week. Muscles biopsies will be taken (i) 12 weeks before commencement of strength training program, (ii) at the beginning of training and (iii) after 12 weeks of strength training. Patients will function as their own controls. Blood samples will be collected simultaneously in order to follow the development of the strength training. Furthermore, participants will be assessed through at number of functional tests and questionnaires evaluating their strength, balance and social/ psychological status.

Subjects are recruited through their association with Odense University Hospital. In the present study, the participants become part of a social network, while participating in organized training sessions, and thus have a possibility to make contact with other ALS patients in the same situation as themselves.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Amyotrophic lateral sclerosis (ALS)

Exclusion Criteria:

* Late stage ALS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Improved muscle strength | 12 weeks
  Measured by Power Rig, KinCom (RFD, Interpolated twich), Calf Press exercises as well as Sway analysis and functional assesments (Timed-up-go + chair rise) Immunohistochemical, genearray, ELISA and Western Blotting analysis techniques are used to gain further data/insight.

SECONDARY OUTCOMES:
Physical, social and mental quality of life | 24 month
  SF-36, Barthel-20, ALSFRS-r and own designed questionaire (physical activity).

CONTACTS AND LOCATIONS:
Overall Officials: Henrik D Schroeder, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Clinical Research, Odense University Hospital, University of Southern Denmark, Odense C, Fyn, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data has been and will be published. Individual participant data may not be available.